CLINICAL TRIAL: NCT04277104
Title: Improving Slow Wave Sleep by Auditory Stimulation to Enhance Memory Consolidation and New Learning in Healthy Older Adults and Older Individuals at Risk for Dementia
Brief Title: Does Acoustic Stimulation During Sleep Boost Slow Wave Sleep and Memory Performance?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2018-01979
Record Dates: First submitted 2020-02-17; First posted 2020-02-20 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Healthy; Mild Cognitive Impairment; Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Healthy intervention (Experimental): Acoustic stimulation
  Interventions: Other: Closed loop acoustic stimulation
- Healthy sham (Sham Comparator): No stimulation
  Interventions: Other: Sham acoustic stimulation
- At risk intervention (Experimental): Acoustic stimulation
  Interventions: Other: Closed loop acoustic stimulation
- At risk sham (Sham Comparator): No stimulation
  Interventions: Other: Sham acoustic stimulation
- MCI (mild cognitive impairment) intervention (Experimental): Acoustic stimulation
  Interventions: Other: Closed loop acoustic stimulation
- MCI (mild cognitive impairment) sham (Sham Comparator): No stimulation
  Interventions: Other: Sham acoustic stimulation

INTERVENTIONS:
Other: Closed loop acoustic stimulation — The intervention consists of three consecutive nights of closed loop acoustic stimulation during slow wave sleep. An established closed-loop algorithm is utilized that detects slow oscillations in the electroencephalogram and is programmed to present short tones (50 ms) into their up-states. Tones will be presented via a headband with integrated speakers. The procedure does not wake participants
  Arms: At risk intervention; Healthy intervention; MCI (mild cognitive impairment) intervention
Other: Sham acoustic stimulation — Sham acoustic stimulation: participants wear the headband but no stimuli are delivered during slow wave sleep. This ensures that in both the control and the intervention group the conscious experiences are the same.
  Arms: At risk sham; Healthy sham; MCI (mild cognitive impairment) sham

SUMMARY:
With aging the amount of slow wave sleep decreases drastically and this disruption is markedly exaggerated in older adults suffering from mild cognitive impairment and Alzheimer's disease. Critically, the disruption of slow wave sleep and cognitive decline seem bidirectionally linked forming a vicious cycle. In the long run, improving slow wave sleep might be a useful intervention tool to delay the onset of cognitive decline. The present study aims at improving slow wave sleep and memory functions through a closed-loop acoustic stimulation approach. A closed-loop algorithm is used that detects slow waves in the electroencephalogram and is programmed to present short tones (50 ms) in the rhythm of these waves. This procedure has shown to boost both slow wave sleep as well as memory performance, mainly in young adults and when applied for one night. Here, the investigators apply tones via multiple consecutive nights and assess memory performance during this 3-night intervention.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Fluent in German
* Normal or corrected to normal vision
* Unimpaired hearing
* For healthy group: Montreal Cognitive Assessment Score ≥ 26
* For MCI group: Montreal Cognitive Assessment Score < 26
* For at risk group: smoker, high cholesterol, high blood pressure and high fasting plasma glucose OR smoker, high BMI, physically inactive, unhealthy dietary habits

Exclusion Criteria:

* Known sleep problems such as Insomnia, restless leg syndrome, apnea
* Irregular sleep pattern
* Symptoms of depression
* History of untreated severe neurological and psychiatric diseases
* Alcohol or substance abuse
* Use of medication acting on the central nervous system

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-10-20 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline episodic memory performance after three nights of intervention | The change in memory performance will be assessed between the baseline measurement (evening before the first intervention night) and on the morning of the last intervention night (1 hour after waking), 3 days after initial encoding
  Face-occupation associative memory task: encoding of 40 faces coupled with 40 occupations takes place on the evening of the first intervention night followed by a retrieval session (BASELINE). Feedback-based retrieval sessions take place on the following mornings and evenings of three consecutive intervention nights (4 feedback-based encoding sessions). After the last intervention night a retrieval session without feedback is performed upon waking (ASSESSMENT OF CHANGE)
Change from baseline performance in computer-based verbal new learning task (episodic memory) after three nights of intervention | The change in new learning performance will be assessed between the baseline measurement (morning before the first intervention night) and on the morning of the last intervention night (1.5 hour after waking), 3 days after.
  Verbal associative memory task: a list of 30 moderately associated word pairs (e.g. balloon-air) are presented on a screen. The respective word pairs are displayed for five seconds each and participants are asked to memorize them. After a one-minute break, a cued recall follows in which one word of each pair is randomly shown and participants are prompted to name the matching second word (BASELINE). After the last intervention night a different list of 30 word pairs is used for another session of encoding and retrieval (ASSESSMENT OF CHANGE)

SECONDARY OUTCOMES:
Improvements in sleep physiology | Three consecutive nights of EEG measurement/polysomnography
  EEG-data: Quality of slow wave sleep, number of slow oscillations, number of sleep spindles can all be measured by the data provided by the electroencephalographic recordings. A high densitiy electrode cap with 128 channels is used for this purpose.
Improvement in episodic memory performance at follow-ups | One week as well as 3 months after intervention
  Face-occupation associative memory task
Improvement in new learning of episodic memory at follow-ups | One week as well as 3 months after intervention
  Verbal associative memory task
Decreases in plasma amyloid-beta | Blood samples will be taken twice: on the morning before the first intervention night, on the morning after the last intervention night (3 days apart)

OTHER OUTCOMES:
General cognitive functions: working memory | Assessed four times: on the morning before the first intervention night, on the morning after the last intervention night, one week after and 3 months after the intervention
  A computer based visual n-back task is performed (established task for working memory)
General cognitive functions: cognitive flexibility | Assessed four times: on the morning before the first intervention night, on the morning after the last intervention night, one week after and 3 months after the intervention
  A computer based task switch task is performed (established task for cognitive flexibility)
General cognitive functions: cognitive inhibition | Assessed four times: on the morning before the first intervention night, on the morning after the last intervention night, one week after and 3 months after the intervention
  A computer based go/no go task is performed (established task for cognitive inhibition)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Klöppel, Prof., Principal Investigator — University hospital of old age psychiatry and psychotherapy
Locations (1):
- University Hospital of Old Age Psychiatry and Psychotherapy, Bern, Switzerland

REFERENCES:
- [Derived] Zeller CJ, Wunderlin M, Wicki K, Teunissen CE, Nissen C, Zust MA, Kloppel S. Multi-night acoustic stimulation is associated with better sleep, amyloid dynamics, and memory in older adults with cognitive impairment. Geroscience. 2024 Dec;46(6):6157-6172. doi: 10.1007/s11357-024-01195-z. Epub 2024 May 14. PMID 38744792